CLINICAL TRIAL: NCT01945983
Title: The Comparison Between Early Norepinephrine Use and Standard Treatment During Severe Sepsis and Septic Shock Resuscitation.
Brief Title: Early Use of Norepinephrine in Septic Shock Resuscitation
Acronym: CENSER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si507/2013
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Septic Shock; Severe Sepsis
Keywords: Septic shock; Severe sepsis; Norepinephrine
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early norepinephrine (Active Comparator): Norepinephrine 4 mg in 5% dextrose water 250 ml Intravenous infusion rate range from 8 to 15 ml/hour, adjusted according to patient's body weight to achieve norepinephrine 0.05microgram/kg/min Continuous drip for 48 hours.
  Interventions: Drug: Early norepinephrine
- Placebo (Placebo Comparator): 5% dextrose water 250 ml Intravenous infusion rate range from 8 to 15 ml/hour. Adjust rate of infusion according to patient's body weight to achieve dosage of norepinephrine comparable to 0.05 microgram/kg/min Continuous drip for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Early norepinephrine — Initiation of norepinephrine, a strong vasoconstrictor, at the initiation of septic shock management, together with fluid resuscitation.
  Other Names: Early vasopressor therapy
  Arms: Early norepinephrine
Drug: Placebo — 5% dextrose water intravenous drip in the same rate of calculated norepinephrine for the patient's body weight
  Other Names: 5%D/W infusion as the placebo of norepinephrine.
  Arms: Placebo

SUMMARY:
Current septic shock guideline recommends fluid resuscitation as the first treatment. Vasopressors, including norepinephrine is recommended to start after achieve adequate fluid therapy. This can cause a certain duration of systemic hypotension before vasopressor is commenced. Initiation of norepinephrine together with fluid therapy soon after diagnosis of septic shock may increase blood pressure quicker than start treatment with intravenous fluid alone. The rapid restoration of perfusion pressure may improve septic shock outcome.

DETAILED DESCRIPTION:
We will include severe infection patient who had evidence of organ dysfunction and hypotension and randomize into 2 groups as following:

1. Control group. The patient will receive treatment according to septic shock guideline 2013, which start with intravenous fluid replacement until achieve target central venous pressure (CVP) or pulmonary capillary wedge pressure (PCWP) or other fluid responsive test goal. If the patient's mean arterial blood pressure still lower than 65 mmHg, then norepinephrine or dopamine will initiate to rise blood pressure. The patient will receive 5% dextrose water as the placebo of norepinephrine.
2. Early norepinephrine group. The patient will receive fluid therapy together with low dose of norepinephrine (0.05 mcg/kg/min). If after titrate intravenous fluid therapy until achieve goal CVP or PCWP or other fluid responsive test, but the mean blood pressure still lower than 65 mmHg, then additional titrate dose of norepinephrine will be given to the patient according to standard septic shock guideline.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Diagnosed severe sepsis or septic shock according to survival sepsis campaign 2013
* Mean arterial pressure < 65 mmHg

Exclusion Criteria:

* Pregnancy
* Severe underlying condition that unexpected to survive more than 48 hours
* Severe peripheral vascular disease
* Patient who required major surgery within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Therapeutic goal achievement | 6 hours
  Therapeutic goal including
  1. Mean arterial blood pressure > or = 65 mmHg
  2. Evidence of adequate tissue perfusion which include continuation of urine output > or = 0.5 ml/kg/hour for 2 hours or decreasing of serum lactate > or = 10 percent in 1 to 2 hours.

SECONDARY OUTCOMES:
Mortality rate | 28 days

OTHER OUTCOMES:
Survive with organ support free days | 28 days
  The days that patient can survive without vasopressor, ventilator support and renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Permpikul, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Result] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Derived] Permpikul C, Tongyoo S, Viarasilpa T, Trainarongsakul T, Chakorn T, Udompanturak S. Early Use of Norepinephrine in Septic Shock Resuscitation (CENSER). A Randomized Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1097-1105. doi: 10.1164/rccm.201806-1034OC. PMID 30704260